CLINICAL TRIAL: NCT02784106
Title: Phase IIa Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of M2951 in Subjects With Rheumatoid Arthritis on Stable Methotrexate Therapy
Brief Title: Safety and Efficacy Study of M2951 in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200527-0081; 2016-000064-42 (EudraCT Number)
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; M2951; Bruton's Tyrosine Kinase (BTK)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — evobrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo: Double-Blind Treatment Period (Placebo Comparator)
  Interventions: Drug: Placebo
- M2951: Double-Blind Treatment Period (Experimental)
  Interventions: Drug: M2951
- Placebo/M2951: Open Label Extension Period (Experimental)
  Interventions: Drug: M2951
- M2951/M2951: Open Label Extension Period (Experimental)
  Interventions: Drug: M2951

INTERVENTIONS:
Drug: Placebo — Participants received placebo matched to M2951 twice daily up to Day 84 during the double-blind treatment period.
  Arms: Placebo: Double-Blind Treatment Period
Drug: M2951 — Participants received 50 milligrams (mg) M2951 orally twice daily up to Day 84 during the double-blind treatment period.
  Other Names: Evobrutinib
  Arms: M2951: Double-Blind Treatment Period
Drug: M2951 — Participants who received placebo matched to M2951 or M2951 in double-blind treatment period, received 50 mg M2951 orally twice daily up to 26-weeks during the open label extension period.
  Other Names: Evobrutinib
  Arms: M2951/M2951: Open Label Extension Period; Placebo/M2951: Open Label Extension Period

SUMMARY:
M2951 is an investigational drug under evaluation for treatment of autoimmune and inflammatory disorders. The purpose of the study is to assess the efficacy of M2951 in participants with rheumatoid arthritis (RA) currently treated with stable dose of methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 75 years of age at the time of informed consent signature
* Confirmed diagnosis of RA according to 2010 American College of Rheumatology (ACR)/The European League Against Rheumatism (EULAR) RA classification criteria of at least 6 months duration
* Positive RF and/or anti-CCP (anti-cyclic citrullinated peptide)
* Persistently active disease defined as greater than equal to (>=) 6 swollen joints (of 66 counted) and >= 6 tender joints (of 68 counted)
* High-sensitivity C-reactive protein (hsCRP) >= 3.6 milligram per liter (mg/L)
* Treatment for >= 12 weeks with 10 to 25 mg/week MTX at a stable dose for at least 4 weeks prior to dosing with the investigational medicinal product (IMP) and maintained throughout the trial
* Women of childbearing potential must use acceptable methods of contraception for 4 weeks prior to randomization, throughout the trial, and for 90 days after the last dose of IMP. For the purposes of this trial
* Females who are postmenopausal (age-related amenorrhea >= 12 consecutive months and increased follicle-stimulating hormone [FSH] greater than (>) 40 milli international units per milliliter [mIU/mL]), or who have undergone hysterectomy or bilateral oophorectomy are exempt from pregnancy testing. If necessary to confirm postmenopausal status, an FSH will be drawn at Screening
* Acceptable contraception is defined as use of either 2 barrier methods (eg, female diaphragm and male condom), or 1 barrier method in conjunction with one of the following: spermicide, an intrauterine device, or hormonal contraceptives (implant or oral)
* Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at Day 1/randomization before dosing.

Exclusion Criteria:

* Use of oral corticosteroids > 10 mg daily prednisone equivalent, use of injectable corticosteroids, or change in dose of corticosteroids within 2 weeks prior to Screening or during Screening
* Initiation or change in dose for nonsteroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to Screening
* Treatment with tofacitinib, other Bruton's Tyrosine Kinase (BTK) inhibitors, or a biologic disease-modifying antirheumatic drug (DMARD; eg, anti-tumor necrosis factor alpha [anti-TNF-α], tocilizumab [anti-interleukin-6 receptor], abatacept [CTLA4-Fc]), or other immunosuppressive drugs(sulfasalazine would be acceptable at a stable dose) other than methotrexate within 3 months prior to Screening or during Screening
* Treatment with anti-CD20 therapy (eg, rituximab) within 12 months prior to Screening or during Screening
* Immunologic disorder other than Rheumatoid Arthritis (RA), with the exception of secondary Sjogren's syndrome associated with RA, and well-controlled diabetes or thyroid disorder, or any other condition requiring oral, intravenous, intramuscular, or intra-articular corticosteroid therapy
* Vaccination with live or live-attenuated virus vaccine within 1 month prior to Screening
* Active, clinically significant, viral, bacterial, or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 4 weeks of Screening or during Screening, or completion of oral anti-infectives within 2 weeks before or during Screening, or a history of recurrent infections (ie, 3 or more of the same type of infection in a 12-month rolling period). Vaginal candidiasis, onychomycosis, and genital or oral herpes simplex virus considered by the Investigator to be sufficiently controlled would not be exclusionary
* History of or positive testing for human immunodeficiency virus (HIV), hepatitis C antibody and/or polymerase chain reaction, hepatitis B surface antigen (HBsAg) (+) and/or hepatitis B core total, and/or IgM antibody (+) at Screening
* History of or current diagnosis of active tuberculosis (TB); undergoing treatment for latent TB infection (LTBI); untreated LTBI (as determined by documented results within 3 months of the Screening Visit of a positive TB skin test with purified protein derivative with induration >= 5 millimeter (mm), a positive QuantiFERON-TB test or positive or borderline T-SPOT [Elispot] test); or positive QuantiFERON-TB test at Screening. Participants with documented completed appropriate LTBI treatment would not be excluded and are not required to be tested
* Participants with current household contacts with active TB will also be excluded
* Indeterminate QuantiFERON-TB or T-SPOT tests may be repeated once, and will be considered positive if retest results are positive or indeterminate
* History of cancer, except adequately treated basal cell or squamous cell carcinomas of the skin (no more than 3 lesions requiring treatment in lifetime) or carcinoma in situ/cervical intraepithelial neoplasia of the uterine cervix, unless considered cured > 5 years
* Clinically significant abnormality on electrocardiogram (ECG), or an active infective process or any other clinically significant abnormality on Screening chest X-ray (CXR) taken within 4 weeks of the first dose, per Investigator opinion. If a CXR has been taken within the previous 3 months and results are available and normal, the CXR does not need to be carried out
* B cell (CD19) count less than (<) 50% of the lower limit of normal at Screening
* Significant cytopenia including absolute neutrophil count < 1,500/ mm^3, platelet count < 100,000/mm^3, or absolute lymphocyte count < 1,000/mm^3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-07-31 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (2):
- U.S. Medical Information, Billerica, Massachusetts, United States
- Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 12-week double-blind treatment period and a 26-week open-label extension period. Primary and secondary outcome measures were planned to be analyzed for double-blind treatment period only.
Groups:
- Placebo: Double-Blind Treatment Period: Participants received placebo matched to M2951 twice daily up to Day 84 during the double-blind treatment period.
- M2951: Double-Blind Treatment Period: Participants received 50 milligrams (mg) M2951 orally twice daily up to Day 84 during the double-blind treatment period.
- Placebo/M2951: Open-Label Extension Period: Participants who received placebo matched to M2951 in double-blind treatment period, received 50 mg M2951 orally twice daily up to 26-weeks during the open-label extension period.
- M2951/M2951: Open-Label Extension Period: Participants who received M2951 in double-blind treatment period, received 50 mg M2951 orally twice daily up to 26-weeks during the open-label extension period.
Period: Double-Blind Treatment Period (12 Weeks)
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period | Placebo/M2951: Open-Label Extension Period | M2951/M2951: Open-Label Extension Period
Started | 32 | 33 | 0 | 0
Completed | 24 | 27 | 0 | 0
Not Completed | 8 | 6 | 0 | 0
Not completed — Adverse Event | 3 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Period: Open-Label Extension Period (26 Weeks)
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period | Placebo/M2951: Open-Label Extension Period | M2951/M2951: Open-Label Extension Period
Started | 0 | 0 | 18 | 21
Completed | 0 | 0 | 15 | 19
Not Completed | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of M2951 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.19) | 53.8 (10.73) | 53.4 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 31 | 32 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieved American College of Rheumatology-20 (ACR20) Response
Description: ACR 20 response: greater than or equal to (>=) 20 percent (%) improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=20% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI); and 5) acute phase reactant as measured by high-sensitivity C-reactive protein (hsCRP). Proportion of ACR20 responders = Number of participants with ACR20 response divided by total participants.
Time Frame: Day 84
Population: The Modified Intent-to-Treat (mITT) Analysis Set included all participants who received at least 1 dose of M2951 or placebo and have at least 1 available ACR20 evaluation at a time point post-dose.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
proportion of participants | 0.42 | 0.52
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Test type: Superiority; Difference in Proportion of Responders = 0.10, 80% CI 2-sided [-0.07 to 0.25]

2. Secondary Outcome: Mean Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP) at Day 28
Description: Mean change in the hsCRP concentration from baseline at Day 28 was reported.
Time Frame: Baseline, Day 28
Population: mITT analysis Set included all participants who received at least 1 dose of M2951 or placebo and have at least 1 available ACR20 evaluation at a time point post-dose.
Measure: Mean (Standard Error); unit: milligram/milliliter (mg/mL)
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
milligram/milliliter (mg/mL) | -0.80 (2.00) | -2.72 (1.93)
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Test type: Superiority; Difference in Mean Changes = -1.93, 80% CI 2-sided [-5.54 to 1.69]

3. Secondary Outcome: Proportion of Participants Achieving American College of Rheumatology-50 (ACR50) Response
Description: ACR 50 response: >=50% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=50% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function measured by HAQ-DI; and 5) acute phase reactant as measured by hsCRP. Proportion of ACR50 responders = Number of participants with ACR50 response divided by total participants.
Time Frame: Day 28, Day 56 and Day 84
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
proportion of participants
  Day 28 | 0.10 | 0.06
  Day 56 | 0.23 | 0.18
  Day 84 | 0.23 | 0.21
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 28; Test type: Superiority; Difference in Proportion of Responders = -0.04, 80% CI 2-sided [-0.13 to 0.06]
Statistical Analysis 2: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 56; Test type: Superiority; Difference in Proportion of Responders = -0.04, 80% CI 2-sided [-0.18 to 0.09]
Statistical Analysis 3: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 84; Test type: Superiority; Difference in Proportion of Responders = -0.01, 80% CI 2-sided [-0.15 to 0.12]

4. Secondary Outcome: Proportion of Participants Achieving American College of Rheumatology-70 (ACR70) Response
Description: ACR 70 response: >=70% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=70% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function measured by HAQ-DI; and 5) acute phase reactant as measured by hsCRP. Proportion of ACR70 responders = Number of participants with ACR70 response divided by total participants.
Time Frame: Day 28, Day 56 and Day 84
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
proportion of participants
  Day 28 | 0.00 | 0.06
  Day 56 | 0.03 | 0.06
  Day 84 | 0.13 | 0.09
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 28; Test type: Superiority; Difference in Proportion of Responders = 0.06, 80% CI 2-sided [0.01 to 0.14]
Statistical Analysis 2: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 56; Test type: Superiority; Difference in Proportion of Responders = 0.03, 80% CI 2-sided [-0.05 to 0.11]
Statistical Analysis 3: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 84; Test type: Superiority; Difference in Proportion of Responders = -0.04, 80% CI 2-sided [-0.15 to 0.07]

5. Secondary Outcome: Mean Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP) at Day 84
Description: Mean change in the hsCRP concentration from baseline at Day 84 was reported.
Time Frame: Baseline, Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/mL
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
mg/mL | -2.14 (2.20) | -3.54 (2.13)
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Test type: Superiority; Difference in Mean Changes = -1.40, 80% CI 2-sided [-5.37 to 2.58]

6. Secondary Outcome: Mean Change From Baseline in Disease Activity Score Based on a 28 Joint Count High-Sensitivity C-Reactive Protein (DAS28-hsCRP) at Day 28 and 84
Description: Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28)+ 0.014* participant's global assessment of disease activity + 0.36*natural log(hsCRP+1) +0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Day 28 and Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
units on a scale
  Change at Day 28 | -0.79 (0.14) | -0.87 (0.13)
  Change at Day 84 | -1.35 (0.20) | -1.28 (0.19)
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 28; Test type: Superiority; Difference in Mean Changes = -0.08, 80% CI 2-sided [-0.33 to 0.16]
Statistical Analysis 2: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Day 84; Test type: Superiority; Difference in Mean Changes = 0.07, 80% CI 2-sided [-0.29 to 0.43]

7. Secondary Outcome: Proportion of Participants With Disease Activity Score- High Sensitivity C-Reactive Protein (DAS28-hsCRP) Value Less Than (<) 3.2
Description: DAS28-hsCRP consisted of composite score of following variables: TJC28, SJC28, hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP =0.56* sqrt(TJC28) + 0.28*sqrt(SJC28)+ 0.014* participant's global assessment of disease activity + 0.36*natural log(hsCRP+1) +0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity. Proportion of participants with DAS28-hsCRP value <3.2 were reported.
Time Frame: Day 84
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
proportion of participants | 0.13 | 0.21
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Test type: Superiority; Difference in Proportion of Participants = 0.08, 80% CI 2-sided [-0.04 to 0.21]

8. Secondary Outcome: Proportion of Participants With Disease Activity Score- High Sensitivity C-Reactive Protein (DAS28-hsCRP) Value Less Than (<) 2.6
Description: DAS28 consisted of composite score of following variables: TJC28, SJC28, hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP =0.56* sqrt (TJC28) + 0.28*sqrt (SJC28)+ 0.014* participant's global assessment of disease activity + 0.36*natural log(hsCRP+1) +0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity. Proportion of participants with DAS28-hsCRP value <2.6 were reported.
Time Frame: Day 84
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
proportion of participants | 0.10 | 0.06
Statistical Analysis 1: Comparison: Placebo: Double-Blind Treatment Period vs M2951: Double-Blind Treatment Period; Test type: Superiority; Difference in Proportion of Participants = -0.04, 80% CI 2-sided [-0.13 to 0.06]

9. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Day 28 and 84
Description: Erythrocyte sedimentation rate (ESR) is a type of blood test that measures how quickly erythrocytes (red blood cells) settle at the bottom of a test tube that contains a blood sample. Higher values indicate inflammation in the body.
Time Frame: Baseline, Day 28 and Day 84
Population: mITT analysis set included all participants who received at least 1 dose of M2951 or placebo and have at least 1 available ACR20 evaluation at a time point post-dose. Here "Number Analyzed" signified those participants who were evaluable for this endpoint at the specified time point.
Measure: Mean (Standard Deviation); unit: millimeter/hour (mm/hour)
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
millimeter/hour (mm/hour)
  Change at Day 28: number analyzed (Participants) | 29 | 32
  Change at Day 28 | -3 (36.9) | -7 (22.1)
  Change at Day 84: number analyzed (Participants) | 25 | 25
  Change at Day 84 | -3 (21.0) | -9 (21.1)

10. Secondary Outcome: Change From Baseline in Anti-cyclic Citrullinated Peptide (Anti-CCP) Antibody Levels at Day 28 and 84
Description: Anti-cyclic citrullinated peptide (anti-CCP) is an antibody present in most rheumatoid arthritis participants.
Time Frame: Baseline, Day 28 and Day 84
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units/milliliter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
units/milliliter
  Change at Day 28: number analyzed (Participants) | 29 | 32
  Change at Day 28 | 168 (991.1) | -138 (720.9)
  Change at Day 84: number analyzed (Participants) | 25 | 25
  Change at Day 84 | 301 (1282.6) | -396 (736.8)

11. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF) at Day 28 and 84
Description: Rheumatoid Factor is an anti-body present in the blood.
Time Frame: Baseline, Day 28 and Day 84
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kiloUnit/Liter (kU/L)
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 31 | 33
kiloUnit/Liter (kU/L)
  Change at Day 28: number analyzed (Participants) | 29 | 32
  Change at Day 28 | -30 (124.2) | -7 (59.7)
  Change at Day 84: number analyzed (Participants) | 25 | 25
  Change at Day 84 | -34 (132.1) | -26 (79.9)

12. Secondary Outcome: Change From Baseline in Global Assessment of Disease Activity Based on Visual Analog Scale (VAS) Score at Day 84
Description: The participant's overall assessment of disease activity was recorded using the 100 millimeter (mm) horizontal visual analog scale (VAS). The scale ranged from 0-100 mm, where 0 indicated no disease activity (symptom free and no arthritis symptoms) and 100 represented maximum disease activity (maximum arthritis disease activity).
Time Frame: Baseline, Day 84
Population: mITT analysis Set included all participants who received at least 1 dose of M2951 or placebo and have at least 1 available ACR20 evaluation at a time point post-dose. Here, "Overall Number of Participants Analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 25 | 26
millimeter | -21 (23.5) | -24 (24.6)

13. Secondary Outcome: Change From Baseline in Self-assessment of Pain Based on Visual Analog Scale (VAS) Score at Day 84
Description: The participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 indicated no pain and 100 indicated worst possible pain.
Time Frame: Baseline, Day 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 25 | 26
millimeter | -19 (21.8) | -22 (22.0)

14. Secondary Outcome: Change From Baseline in Self-assessment of Disability Using Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Day 84
Description: The HAQ-DI questionnaire assessed the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Day 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 25 | 26
units on a scale | -0.3 (0.44) | -0.3 (0.41)

15. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity Scale Based on Visual Analog Scale (VAS) Score at Day 84
Description: The Physician's Global Assessment of Disease Activity was recorded using the 100 mm horizontal VAS. Physician rated participant's arthritis disease activity on a scale ranged from 0-100 mm, where 0 indicated no disease activity (no arthritis) and 100 represented maximum disease activity (maximum arthritis).
Time Frame: Baseline, Day 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 25 | 26
millimeter | -33 (20.3) | -30 (22.7)

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 16 Weeks
Population: The Safety Analysis Set included all participants who received at least 1 dose of M2951 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 32 | 33
Participants
  TEAEs | 16 | 22
  SAEs | 0 | 1

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity
Description: Grade 3 and 4 TEAES as per National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03 (NCI-CTCAE v 4.03) were presented. Grade 3 refers to severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care and Activity of daily living (ADL).Grade 4 refers to Life-threatening consequences; where urgent intervention indicated.
Time Frame: Baseline up to 16 Weeks
Population: The Safety Analysis Set included all participants who received at least 1 dose of M2951 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 32 | 33
Participants
  NCI-CTCAE Severity grade >=3 | 2 | 3
  NCI-CTCAE Severity grade >=4 | 0 | 1

18. Secondary Outcome: Number of Participants With Grade 3 or Higher Clinically Significant Abnormality for Hematology, Biochemistry, Urinalysis or Coagulation
Description: Clinically significant abnormalities for hematology, biochemistry or coagulation were graded with National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 toxicity grades, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = death. Participants with grade 3 or higher were reported.
Time Frame: Baseline up to 16 Weeks
Population: The Safety Analysis Set included all participants who received at least 1 dose of M2951 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 32 | 33
Participants
  Hematology | 2 | 0
  Biochemistry | 4 | 2
  Coagulation | 0 | 0
  Urinalysis | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital sign assessment included blood pressure, pulse rate, respiratory rate and temperature. Clinical significance was determined by the investigator.
Time Frame: Baseline up to 16 Weeks
Population: The Safety Analysis Set included all participants who received at least 1 dose of M2951 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 32 | 33
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings
Description: The 12-lead ECG recordings were obtained after 10 minutes of rest in a semi-supine position. The ECG parameters obtained directly from the computerized 12-lead ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, and QT interval. Clinical significance was determined by the investigator.
Time Frame: Baseline up to 16 Weeks
Population: The Safety Analysis Set included all participants who received at least 1 dose of M2951 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 32 | 33
Participants | 0 | 0

21. Secondary Outcome: Plasma Concentration of M2951
Time Frame: Pre-dose at Day 1; 0.25, 0.5, 1.0, 2.0, 4.0, 6.0 hours post-dose at Day 1 and Day 29
Population: The Pharmacokinetic (PK) Analysis Set included all participants who receive at least 1 dose of M2951 and have at least 1 quantifiable M2951 plasma concentration at a scheduled PK time point post-dose. Here "Number Analyzed" signified those participants who were evaluable for this endpoint at the specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 33
nanogram per milliliter (ng/mL)
  Day 1: Pre-Dose: | 0.00 (NA) — Statistical Analysis was not applicable as mean concentration of the drug is zero.
  Day 1: 0.25 hours post-dose | 10.3 (23.37)
  Day 1: 0.5 hours post-dose | 80.5 (136.9)
  Day 1: 1 hour post-dose | 160 (219.7)
  Day 1: 2 hours post-dose | 125 (111.9)
  Day 1: 4 hours post-dose | 47.3 (41.62)
  Day 1: 6 hours post-dose | 23.7 (20.92)
  Day 29: 0.25 hours post-dose: number analyzed (Participants) | 28
  Day 29: 0.25 hours post-dose | 22.0 (71.57)
  Day 29: 0.5 hours post-dose: number analyzed (Participants) | 28
  Day 29: 0.5 hours post-dose | 88.4 (114.1)
  Day 29: 1 hour post-dose: number analyzed (Participants) | 28
  Day 29: 1 hour post-dose | 120 (107.2)
  Day 29: 2 hours post-dose: number analyzed (Participants) | 27
  Day 29: 2 hours post-dose | 82.3 (53.82)
  Day 29: 4 hours post-dose: number analyzed (Participants) | 28
  Day 29: 4 hours post-dose | 62.1 (82.39)
  Day 29: 6 hour post-dose: number analyzed (Participants) | 27
  Day 29: 6 hour post-dose | 37.2 (43.96)

22. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 6 Hours (AUC 0-6h) of M2951
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0 hours post-dose at Day 1 and Day 29
Population: PK Analysis Set included all participants who receive at least 1 dose of M2951 and have at least 1 quantifiable M2951 plasma concentration at a scheduled PK time point post-dose. Here "Number Analyzed" signified those participants who were evaluable for this endpoint at the specified time point.
Measure: Mean (Standard Deviation); unit: hours*nanogram/milliliter
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 33
hours*nanogram/milliliter
  Day 1 | 431 (390.9)
  Day 29: number analyzed (Participants) | 26
  Day 29 | 414 (268.4)

23. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of M2951
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0 hours post-dose at Day 1 and Day 29
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 33
ng/mL
  Day 1 | 206 (214.7)
  Day 29: number analyzed (Participants) | 27
  Day 29 | 171 (130.1)

24. Secondary Outcome: Plasma Concentration Observed Immediately Before Dosing on Day 29 (Cpre) of M2951
Time Frame: Pre-dose on Day 29
Population: PK Analysis Set included all participants who receive at least 1 dose of M2951 and have at least 1 quantifiable M2951 plasma concentration at a scheduled PK time point post-dose. Here, "Overall Number of Participants Analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 28
ng/mL | 5.47 (4.735)

25. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of M2951
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0 hours post-dose at Day 1 and Day 29
Population: as for outcome 22
Measure: Median (Full Range); unit: hour
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 33
hour
  Day 1 | 1.00 [0.50 to 4.00]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 1.00 [0.50 to 6.00]

26. Secondary Outcome: Accumulation Ratio for Area Under the Concentration-Time Curve From Time Zero to 6 Hours (Racc [AUC0-6h]) of M2951
Description: Accumulation ratio for AUC was calculated as AUC 0-6h, Day 29 divided by AUC 0-6h, Day 1
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0 hours post-dose at Day 1 and Day 29
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 26
ratio | 1.38 (1.134)

27. Secondary Outcome: Accumulation Ratio for Observed Maximum Plasma Concentration (Racc [Cmax]) of M2951
Description: Accumulation ratio for Cmax , was calculated as Cmax, Day 29 divided by Cmax, Day1
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 2.0, 4.0, 6.0 hours post-dose at Day 1 and Day 29
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 27
ratio | 1.52 (1.929)

28. Secondary Outcome: Absolute Immunoglobulin Levels at Day 85
Description: Following immunoglobulin levels were measured: Immunoglobulin A , Immunoglobulin G, Immunoglobulin G Subclass 1, Immunoglobulin G Subclass 2, Immunoglobulin G Subclass 3, Immunoglobulin G Subclass 4, Immunoglobulin M.
Time Frame: Baseline, Day 85
Population: PD Analysis Set included all participants who received at least 1 dose of M2951 or placebo and have at least 1 measured PD endpoint, not including BTK occupancy, at a scheduled PD time point post-dose. Here, "Overall Number of Participants Analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: gram/Liter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 10 | 12
gram/Liter
  Immunoglobulin A | 2.09 (0.968) | 2.77 (1.323)
  Immunoglobulin G | 10.61 (3.897) | 9.88 (2.498)
  Immunoglobulin G Subclass 1 | 6.20 (2.338) | 5.41 (1.574)
  Immunoglobulin G Subclass 2 | 3.59 (1.644) | 3.74 (1.205)
  Immunoglobulin G Subclass 3 | 1.05 (0.551) | 0.93 (0.510)
  Immunoglobulin G Subclass 4 | 0.394 (0.2474) | 0.684 (0.6286)
  Immunoglobulin M | 1.16 (0.365) | 1.16 (0.642)

29. Secondary Outcome: Absolute Change From Baseline in Immunoglobulin Levels at Day 85
Description: as for outcome 28
Time Frame: Baseline, Day 85
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: gram/Liter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 10 | 12
gram/Liter
  Immunoglobulin A | -0.07 (0.263) | -0.04 (0.133)
  Immunoglobulin G | 0.02 (1.281) | -0.30 (0.517)
  Immunoglobulin G Subclass 1 | 0.11 (0.857) | -0.15 (0.410)
  Immunoglobulin G Subclass 2 | -0.13 (0.477) | -0.17 (0.404)
  Immunoglobulin G Subclass 3 | 0.07 (0.214) | -0.04 (0.209)
  Immunoglobulin G Subclass 4 | -0.028 (0.1073) | -0.046 (0.2576)
  Immunoglobulin M | -0.04 (0.177) | -0.25 (0.255)

30. Secondary Outcome: Absolute B-Cell Levels at Day 85
Time Frame: Day 85
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: cells per micro-liter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 12 | 12
cells per micro-liter | 243 (265.0) | 204 (154.0)

31. Secondary Outcome: Absolute Change From Baseline in B-cell Levels at Day 85
Time Frame: Baseline, Day 85
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: cells per micro-liter
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period
Number analyzed (Participants) | 12 | 12
cells per micro-liter | 76 (242.0) | 11 (73.2)

ADVERSE EVENTS:
Time Frame: Double-Blind Period: Baseline up to 16 weeks; Open-Label Period: Baseline up to 30 weeks
Description: MedDRA version for the double-blind treatment period is version 20.0 and MedDRA version for the open-label extension period is version 20.1
Arm/Group | Placebo: Double-Blind Treatment Period | M2951: Double-Blind Treatment Period | Placebo/M2951: Open-Label Extension Period | M2951/M2951: Open-Label Extension Period
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/33 | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 13/32 | 17/33 | 8/18 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Double-Blind Treatment Period (N=32) | M2951: Double-Blind Treatment Period (N=33) | Placebo/M2951: Open-Label Extension Period (N=18) | M2951/M2951: Open-Label Extension Period (N=21)
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo CNS origin (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Double-Blind Treatment Period (N=32) | M2951: Double-Blind Treatment Period (N=33) | Placebo/M2951: Open-Label Extension Period (N=18) | M2951/M2951: Open-Label Extension Period (N=21)
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 4 | 3 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 3
Lipase increased (Investigations) | 2 | 3 | 0 | 0
Blood glucose increased (Investigations) | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 1 | 0
Amylase increased (Investigations) | 3 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT02784106/SAP_001.pdf
  • Study Protocol (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT02784106/Prot_002.pdf